CLINICAL TRIAL: NCT05791435
Title: Respiratory Biofeedback Sensor for Yoga Practice for Youth With Chronic Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Tariq Rahman, Principal Research Engineer, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1904079; 3R41AT012155-01S1 (NIH)
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback group (Experimental): This group will receive biofeedback to assist with breathing
  Interventions: Device: PneuRIP; Other: biofeedback to assist with breathing
- Non-Biofeedback group (Experimental): This group will only have their breathing monitored after instruction
  Interventions: Device: PneuRIP

INTERVENTIONS:
Device: PneuRIP — Measuring respiratory indices through Respiratory Inductance Plethysmography
  Other Names: Non-invasive breathing monitor
Other: biofeedback to assist with breathing — Measuring respiratory indices through Respiratory Inductance Plethysmography and providing visual biofeedback on a tablet screen
  Arms: Biofeedback group

SUMMARY:
This project will develop and test a wearable breathing monitor that will measure the synchrony in breathing between the diaphragm and chest of children with a pain diagnosis while receiving yoga therapy. Specifically, we will develop a biofeedback system to help improve breathing in pain patients.

DETAILED DESCRIPTION:
This Small Business Technology Transfer (STTR) Phase I application proposes the development and trial of a novel non-invasive real-time breathing sensor - pneuRIP- to show the beneficial effects of respiratory biofeedback on yoga. PneuRIP will be employed to monitor and improve asana (posture) and pranayama (breathing) in yoga in youth with chronic pain. The sensor consists of two inductive bands worn around the chest and abdomen that measure and differentiate diaphragmatic and chest breathing through Respiratory Inductance Plethysmography (RIP). Readings are recorded and analyzed on a small chest-worn unit and wirelessly transmitted to an iPad. Measures include the phase angle between the chest and abdomen; percentage breathing through the ribcage; respiratory rate; and labored breathing index. This sensor takes little time to set up and readings are provided instantaneously.

The first part of the proposal will develop the biofeedback software. The biofeedback component will be related to the synchrony between diaphragmatic and chest breathing, and the relative depth of breathing. This information will be presented to the user visually on an iPad screen in the form of 2 moving bars - one corresponding to the chest and one to the belly.

In the second part of the study, we will test the pneuRIP with biofeedback with 20 youth with pain enrolled in an interdisciplinary pediatric chronic pain program in a large pediatric hospital receiving yoga as one of the therapies. The yoga regimen is 8 sessions, once per week. Subjects will be randomized into two groups: one receiving instruction only on synchronous breathing; the second group will receive biofeedback in addition. Outcome will phase angle between abdomen and ribcage (recorded during each session). Outcomes will inform the feasibility of using real-time biofeedback in yoga with a non-invasive respiratory monitor.

ELIGIBILITY:
Inclusion Criteria:

* Youth with Chronic pain Prescribed yoga therapy as part of treatment plan

Exclusion Criteria:

* Otherwise healthy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours/A.I. duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited in Medical clinic. Dates are 5/1/23-8/29/23
Period: Overall Study
Arm/Group | Biofeedback Group | Non-Biofeedback Group
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofeedback Group | Non-Biofeedback Group | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.14 (2.79) | 16.57 (1.27) | 15.36 (2.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase Angle
Description: Measures synchrony between chest and stomach. The phase angle is measured in degrees. If the chest and stomach move together then the phase angle is zero degrees. If they were to move in opposite directions the phase angle would be 180 degrees.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Biofeedback Group | Non-Biofeedback Group
Number analyzed (Participants) | 7 | 7
degrees | 58 (13.65) | 41 (12.17)

ADVERSE EVENTS:
Time Frame: 4 months
Description: The risk for serious adverse events, non-serious adverse events and all-cause mortality is zero as the study monitored subjects' breathing while performing routine therapy
Arm/Group | Biofeedback Group | Non-Biofeedback Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT05791435/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT05791435/SAP_001.pdf